CLINICAL TRIAL: NCT03289546
Title: Exploring Synergistic Effects Of Aerobic Exercise And Mindfulness Training On Cognitive Function In Older Adults: A Pilot, Proof Of Concept Study
Brief Title: The Active Mind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Elena Salmoirago-Blotcher, Assistant professor of Medicine, The Miriam Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 201602917
Record Dates: First submitted 2017-03-23; First posted 2017-09-21 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Impairment; Cardiovascular Risk Factor
Keywords: mindfulness; exercise; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness training only (Experimental): 1 mindfulness training class (1 hour) every week for 8 weeks.
  Interventions: Behavioral: Mindfulness training
- Aerobic training only (Experimental): 3 aerobic training sessions (1 hour) per week for 12 weeks.
  Interventions: Behavioral: Aerobic training
- mindfulness + aerobic training (Experimental): 2 aerobic training sessions + 1 mindfulness training class every week for 8 weeks, then continue with 3 aerobic training sessions/ week for 4 additional weeks.
  Interventions: Behavioral: Mindfulness training; Behavioral: Aerobic training
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness training — The mindfulness training protocol will include the following basic components of traditional mindfulness-based stress reduction training: 1) training in awareness of sensations ("body scan"); 2) training in the awareness of the sensations of breathing; 3) training in directing the attention to simple activities of daily life, and in recognizing when the attention is no longer focused on a specific object of attention; and 4) training in 'open awareness'.
  Arms: Mindfulness training only; mindfulness + aerobic training
Behavioral: Aerobic training — Exercise sessions will be led by CPR- and exercise-certified YMCA instructors and supervised by the senior research assistant. Sessions will consist of 10 minutes of warm-up, 40 minutes of aerobic exercise (walking on a treadmill), 10 minutes of cool down and stretching. Participants will receive heart monitors at the beginning of the study and will be trained by the senior research assistant to exercise targeting heart rates at 65-75% of the age predicted max heart rate or at an intensity of 12-13 in the Borg scale of the rate of perceived exertion.
  Arms: Aerobic training only; mindfulness + aerobic training

SUMMARY:
The purpose of this study is to explore whether physical exercise, mindfulness training, or both interventions together can improve cognitive function in individuals with multiple risk factors for the development of dementia in the future.

DETAILED DESCRIPTION:
The investigators will test the feasibility and acceptability of a combined mindfulness training + aerobic training intervention, vs. either alone or none to improve cognitive function in older adults with cognitive impairment. The investigators will also obtain estimates of effect sizes (and confidence intervals) on cognitive function. Preliminary analyses will be conducted to explore the mediating role of changes in aerobic capacity, physical activity, vascular risk factors, and mindfulness skills. Assessments will be conducted at baseline, 3-, and 6- months since baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55
2. Being physically inactive (defined as not meeting current AHA recommendations for physical activity, i.e., < 150 min of moderate-intensity aerobic activity per week OR < 75 minutes of vigorous aerobic activity per week
3. Cognitive complaint defined as answering yes to the question "do you feel that your memory or thinking skills have gotten worse recently?"
4. Fluency in English language

Exclusion Criteria:

1. Unwillingness/inability to provide informed consent
2. Contraindications to physical activity as per the participant's PCP assessment
3. Blood pressure >200/110
4. Severe depressive symptoms (defined as Hospital Anxiety and Depression Scale [HADS] depression subscale scores >14)
5. Acute psychosis (from medical record)
6. Severe cognitive impairment (Mini-Mental State Examination [MMSE] score <24)
7. Recent hospitalization (< 6 weeks)
8. Current (at least once a month) mind/body practice (i.e., mindfulness meditation, yoga, or tai chi)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Retention rates of 80% at the final follow-up visit | 3 months from baseline
  The investigators will consider the study feasible under this condition
Number of participants who attended at least 70% of the planned sessions | 3 months from baseline
  The investigators will consider the study feasible under this condition
Number of participants who completed 70% of the assigned individual home practice exercises | 3 months from baseline
  The investigators will consider the study feasible under this condition
Acceptability will be assessed using a satisfaction survey | 3 months from baseline
  Acceptability will be assessed using a satisfaction survey. The intervention will be considered acceptable if ≥80% of participants responds that they are at least somewhat satisfied with the intervention.

SECONDARY OUTCOMES:
Effect size on cognitive function | baseline, 3, 6 months
  Preliminary estimates of effect size of mindfulness training alone vs. aerobic training alone, both, or neither on changes from baseline cognitive function.
An exploratory outcome: Mindfulness will be assessed using the Five Facets of Mindfulness questionnaire (short form) | baseline, 3, 6 months
  Five Facets of Mindfulness questionnaire (short form) is a 12-item questionnaire that measures the five identified components of mindfulness meditation: observing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
An exploratory outcome: Depression will be assessed using the Hospital Anxiety and Depression Scale (HADS) | baseline, 3, 6 months
  The HADS is a self-administered questionnaire with two sub-scales (0-21) measuring anxiety and depression, with higher scores indicating greater psychological morbidity
Exploratory outcome: waist-to-hip ratio | baseline, 3, 6 months
  waist-to-hip ratio
An exploratory outcome: Exercise capacity will be assessed via the 6 minute walking test | baseline, 3, 6 months
  The 6 minute walking test
Exploratory outcome: blood pressure | baseline, 3, 6 months
  blood pressure
An exploratory outcome: Social support will be assessed using the Multidimensional Scale of Perceived Social Support | baseline, 3, 6 months
  A 12-item, uni-dimensional tool to measure how one perceives their social support system, including individuals sources of social support (i.e., family, friends, and significant other).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salmoirago-Blotcher, PhD, MD, Principal Investigator — The Miriam Hospital & Warren Alpert Medical School at Brown University
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salmoirago-Blotcher E, DeCosta J, Harris K, Breault C, Dunsiger S, Santos C, Snyder P. Exploring synergistic effects of aerobic exercise and mindfulness training on cognitive function in older adults: Protocol for a pilot randomized controlled trial. Medicine (Baltimore). 2018 May;97(21):e10626. doi: 10.1097/MD.0000000000010626. PMID 29794738